CLINICAL TRIAL: NCT05949320
Title: "Health in Mobile" - The e-Motivational-Interviewing Intervention for Community-dwelling Individuals With Chronic Diseases
Brief Title: "Health in Mobile" for Community-dwelling Individuals With Chronic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: The Hong Kong Society for Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HKSR T591
Record Dates: First submitted 2023-06-29; First posted 2023-07-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Intervention; Control Group
Keywords: Motivational Interviewing; Hypertension; Diabetes Mellitus; Mobile Phone-Based Intervention; mHealth
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- e-MI intervention group (Experimental): 1200 participations are randomized to the e-MI group. They are asked to download the e-MI app and exposed to the related content for 90 days.
  Interventions: Other: e-Motivational Interviewing
- Waiting list control group (No Intervention): 400 participants are randomized to the waiting list control group. They will commence the e-MI intervention after the completion of the e-MI group.

INTERVENTIONS:
Other: e-Motivational Interviewing — This study evaluates a 90-day mobile phone-based intervention using the e-Motivational Interviewing app for individuals with chronic conditions like hypertension and diabetes. The app provides short conversations with health messages and reflective questions on lifestyle choices, such as physical activity and diet. The intervention incorporates "change talk" from Motivational Interviewing and principles from Basic Psychological Needs Theory (BPNT) to encourage positive behavior change. Users interact via multiple-choice questions, promoting self-assessment and reflection. The goal is to facilitate sustained lifestyle changes and improved health outcomes.
  Arms: e-MI intervention group

SUMMARY:
This study aims to provide a mobile-apps-based intervention to facilitate individuals with chronic diseases such as high blood pressure and diabetes to adopt healthy behaviours. The intervention is based on Motivational Interviewing, a clinical technique used to enhance an individual's behavioural changes. The proposed research project comprises developing and validating the "Health in Mobile" app, which we call e-MI, which will then be launched to members of the three District Health Centre Express (DCHEs) who have presented with clinical/preclinical chronic health issues such as high blood pressure and diabetes. The participants are registered members of the three DCHEs. The targeted sample size is 1600 members, with 1200 are in the e-MI group while the other 400 are in the waiting list control group.

DETAILED DESCRIPTION:
Motivational interviewing (MI) is a clinical technique used to enhance an individual's behavioral changes. The MI intervention shares a similar basis as the cognitive behavioral therapy based on the Stages of Change. It has been found effective for enabling individuals to tackle their problems in weight control, substance abuse, and smoking.

The proposed study focuses on facilitating individuals with chronic diseases such as high blood pressure and diabetes to adopt health behaviors. The technique employed to facilitate the behavioral changes is the MI. Previous literature has reported the positive effects of MI in patients with chronic diseases. For instance, promoting weight loss in overweight and obese individuals, improving physical activity self-management in adults with type II diabetes, and regulation in blood pressure level among hypertensive individuals. However, the applications of the MI are mostly via the face-to-face method. Other application methods such as telephone coaching, online synchronous chat and mobile app are delivered as the alternative for communication. Individuals are engaged to enhance or modify certain behaviors via such as instant text interaction with psychologists, messages generated from a predefined system, and messages from interactive tools based on one's situation. Positive intervention effects were observed in these alternative forms of MI in terms of successful weight loss from a mobile app and telephone coaching and smoking cessation from telephone coaching. However, drawbacks include decreased attendance and engagement for lengthy programs, technical issues in delivering messages, and over-simplification of materials. The purpose of this study, therefore, is to deliver the MI to the participants with the use of perceptual learning theories, and the differential focuses on the cognitive and affective components when viewing simple MI messages via an app, and we name it the e-MI.

ELIGIBILITY:
Inclusion Criteria:

* 1) pass the cognitive screening test indicating low risk of mild cognitive impairment and depressive moods;
* 2) age 45 to 75 years;
* 3) completed primary school education or above;
* 4) has a considerate level of information literacy access to mobile phones and tablets;
* 5) agree to participate in the study and provide informed consent.

Exclusion Criteria:

* 1) participants with type 1 diabetes, impaired glucose tolerance, metabolic syndrome, maturity-onset diabetes of youth, or gestational diabetes;
* 2) clinical diagnosis of cardiovascular disease, kidney disease, liver disease, malignant tumour, or new-onset diabetes after organ transplant;
* 3) participants with a psychiatric or neurological disability

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The Chinese Affect Scale | Baseline
  The 12-item Chinese Affect Scale measures positive emotions and negative emotions of the day following each daily e-MI message delivery. Six items assess positive emotions and negative emotions, respectively (Hou et al., 2016). Participants will use a 11-point scale (0=very slightly or not at all, 5=moderately, 10=very much) to indicate the extent to which they were experiencing each emotional state at a sampling moment.
The Chinese Affect Scale | 3 months
  The 12-item Chinese Affect Scale measures positive emotions and negative emotions of the day following each daily e-MI message delivery. Six items assess positive emotions and negative emotions, respectively (Hou et al., 2016). Participants will use a 11-point scale (0=very slightly or not at all, 5=moderately, 10=very much) to indicate the extent to which they were experiencing each emotional state at a sampling moment.
The Chinese Affect Scale | 9 months
  The 12-item Chinese Affect Scale measures positive emotions and negative emotions of the day following each daily e-MI message delivery. Six items assess positive emotions and negative emotions, respectively (Hou et al., 2016). Participants will use a 11-point scale (0=very slightly or not at all, 5=moderately, 10=very much) to indicate the extent to which they were experiencing each emotional state at a sampling moment.
The Chinese version of University of Rhode Island Change Assessment | Baseline
  The Chinese version of University of Rhode Island Change Assessment is a 32-item questionnaire to measure individuals' readiness for health-related changes for positive health-related behaviours.
  The Chinese version of University of Rhode Island Change Assessment comprises 32 items that measure four stages of change. Participants rate each item on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).To calculate the scores for each stage, sum the item scores for the corresponding items in each stage and divide by the number of items in that stage. This will provide an average score for each stage of change. Higher scores indicate a greater readiness for change at that specific stage.
The Chinese version of University of Rhode Island Change Assessment | 3 months
  The Chinese version of University of Rhode Island Change Assessment is a 32-item questionnaire to measure individuals' readiness for health-related changes for positive health-related behaviours.
  The Chinese version of University of Rhode Island Change Assessment comprises 32 items that measure four stages of change. Participants rate each item on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).To calculate the scores for each stage, sum the item scores for the corresponding items in each stage and divide by the number of items in that stage. This will provide an average score for each stage of change. Higher scores indicate a greater readiness for change at that specific stage.
The Chinese version of University of Rhode Island Change Assessment | 9 months
  The Chinese version of University of Rhode Island Change Assessment is a 32-item questionnaire to measure individuals' readiness for health-related changes for positive health-related behaviours.
  The Chinese version of University of Rhode Island Change Assessment comprises 32 items that measure four stages of change. Participants rate each item on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).To calculate the scores for each stage, sum the item scores for the corresponding items in each stage and divide by the number of items in that stage. This will provide an average score for each stage of change. Higher scores indicate a greater readiness for change at that specific stage.
The International Physical Activity Questionnaire - Short Form | Baseline
  The International Physical Activity Questionnaire - Short Form measures participants' intensity and duration of physical activity in their daily lives, covering vigorous-intensity activities, moderate-intensity activities, walking, and sitting time.
The International Physical Activity Questionnaire - Short Form | 3 months
  The International Physical Activity Questionnaire - Short Form measures participants' intensity and duration of physical activity in their daily lives, covering vigorous-intensity activities, moderate-intensity activities, walking, and sitting time.
The International Physical Activity Questionnaire - Short Form | 9 months
  The International Physical Activity Questionnaire - Short Form measures participants' intensity and duration of physical activity in their daily lives, covering vigorous-intensity activities, moderate-intensity activities, walking, and sitting time.
The standard 12-Item Short Form Health Survey | Baseline
  The SF-12 measures eight health domains, which can be grouped into two summary scores: Physical Component Summary (PCS) & Mental Component Summary (MCS).
  Participants are asked to respond to each item considering their health status over the past four weeks. The response options vary depending on the item, with some questions having binary (yes/no) answers, and others using ordinal scales.
  Each of the eight health domains is scored separately, with higher scores indicating better health. The scores for each domain are then standardized and weighted to calculate the PCS and MCS scores. Higher scores on the PCS and MCS represent better health-related quality of life.
The standard 12-Item Short Form Health Survey | 3 months
  The SF-12 measures eight health domains, which can be grouped into two summary scores: Physical Component Summary (PCS) & Mental Component Summary (MCS).
  Participants are asked to respond to each item considering their health status over the past four weeks. The response options vary depending on the item, with some questions having binary (yes/no) answers, and others using ordinal scales.
  Each of the eight health domains is scored separately, with higher scores indicating better health. The scores for each domain are then standardized and weighted to calculate the PCS and MCS scores. Higher scores on the PCS and MCS represent better health-related quality of life.
The standard 12-Item Short Form Health Survey | 9 months
  The SF-12 measures eight health domains, which can be grouped into two summary scores: Physical Component Summary (PCS) & Mental Component Summary (MCS).
  Participants are asked to respond to each item considering their health status over the past four weeks. The response options vary depending on the item, with some questions having binary (yes/no) answers, and others using ordinal scales.
  Each of the eight health domains is scored separately, with higher scores indicating better health. The scores for each domain are then standardized and weighted to calculate the PCS and MCS scores. Higher scores on the PCS and MCS represent better health-related quality of life.
The Treatment Self-Regulation Questionnaire | Baseline
  The 15-item Treatment Self-Regulation Questionnaire will be used to assess the participants' motivation to perform health behaviors in terms of autonomous (intrinsically motivated) versus controlled (extrinsically motivated) over the past two weeks. Responses will range from 1 to 7 for each item (1=not at all true, 4=somewhat true, 7=very true) and will then be averaged to form the score for each self-regulation style (i.e., intrinsic vs. extrinsic).
The Treatment Self-Regulation Questionnaire | 3 months
  The 15-item Treatment Self-Regulation Questionnaire will be used to assess the participants' motivation to perform health behaviors in terms of autonomous (intrinsically motivated) versus controlled (extrinsically motivated) over the past two weeks. Responses will range from 1 to 7 for each item (1=not at all true, 4=somewhat true, 7=very true) and will then be averaged to form the score for each self-regulation style (i.e., intrinsic vs. extrinsic).
The Treatment Self-Regulation Questionnaire | 9 months
  The 15-item Treatment Self-Regulation Questionnaire will be used to assess the participants' motivation to perform health behaviors in terms of autonomous (intrinsically motivated) versus controlled (extrinsically motivated) over the past two weeks. Responses will range from 1 to 7 for each item (1=not at all true, 4=somewhat true, 7=very true) and will then be averaged to form the score for each self-regulation style (i.e., intrinsic vs. extrinsic).
The Contemplation Ladder | Baseline
  The Contemplation Ladder is a visual analog scale designed as a ladder with 11 rungs, numbered from 0 to 10. Each rung represents a different level of readiness to change, ranging from no intention to change (0) to taking action to change (10).
The Contemplation Ladder | 3 months
  The Contemplation Ladder is a visual analog scale designed as a ladder with 11 rungs, numbered from 0 to 10. Each rung represents a different level of readiness to change, ranging from no intention to change (0) to taking action to change (10).
The Contemplation Ladder | 9 months
  The Contemplation Ladder is a visual analog scale designed as a ladder with 11 rungs, numbered from 0 to 10. Each rung represents a different level of readiness to change, ranging from no intention to change (0) to taking action to change (10).
The Chinese version of the 7-item Generalized Anxiety Disorder scale | Baseline
  The Chinese version of the 7-item Generalized Anxiety Disorder scale will be used to assess anxiety symptoms in the past two weeks. Summed scores range from 0 to 21 (0 = not at all, 1 = on several days, 2 = on more than half of the days, 3 = nearly every day). Higher scores indicated greater severity of anxiety symptoms.
The Chinese version of the 7-item Generalized Anxiety Disorder scale | 3 months
  The Chinese version of the 7-item Generalized Anxiety Disorder scale will be used to assess anxiety symptoms in the past two weeks. Summed scores range from 0 to 21 (0 = not at all, 1 = on several days, 2 = on more than half of the days, 3 = nearly every day). Higher scores indicated greater severity of anxiety symptoms.
The Chinese version of the 7-item Generalized Anxiety Disorder scale | 9 months
  The Chinese version of the 7-item Generalized Anxiety Disorder scale will be used to assess anxiety symptoms in the past two weeks. Summed scores range from 0 to 21 (0 = not at all, 1 = on several days, 2 = on more than half of the days, 3 = nearly every day). Higher scores indicated greater severity of anxiety symptoms.
Health Promotion Lifestyle Profile - II: Chinese version Short Form | Baseline
  Health Promotion Lifestyle Profile - II: Chinese version Short Form is a 30-item measure designed for reflecting health promotion lifestyle behaviors. Participants are asked to rate each item on a 4-point Likert scale, ranging from 1 (never) to 4 (routinely). To calculate the scores for each dimension, sum the item scores for the corresponding items in each dimension and divide by the number of items in that dimension. This will provide an average score for each dimension. Higher scores indicate better health-promoting behavior in that specific domain.
Health Promotion Lifestyle Profile - II: Chinese version Short Form | 3 months
  Health Promotion Lifestyle Profile - II: Chinese version Short Form is a 30-item measure designed for reflecting health promotion lifestyle behaviors. Participants are asked to rate each item on a 4-point Likert scale, ranging from 1 (never) to 4 (routinely). To calculate the scores for each dimension, sum the item scores for the corresponding items in each dimension and divide by the number of items in that dimension. This will provide an average score for each dimension. Higher scores indicate better health-promoting behavior in that specific domain.
Health Promotion Lifestyle Profile - II: Chinese version Short Form | 9 months
  Health Promotion Lifestyle Profile - II: Chinese version Short Form is a 30-item measure designed for reflecting health promotion lifestyle behaviors. Participants are asked to rate each item on a 4-point Likert scale, ranging from 1 (never) to 4 (routinely). To calculate the scores for each dimension, sum the item scores for the corresponding items in each dimension and divide by the number of items in that dimension. This will provide an average score for each dimension. Higher scores indicate better health-promoting behavior in that specific domain.
Self-Reported Chronic Medical Conditions | Baseline
  Participants will report whether or not they currently have a list of chronic medical conditions, including but not limited to arthritis, hypertension, heart attack, chronic lung disease, stroke, diabetes, bladder disease, nephrolith, visual problems, hearing problems, and hemorrhoids.
Self-Reported Chronic Medical Conditions | 3 months
  Participants will report whether or not they currently have a list of chronic medical conditions, including but not limited to arthritis, hypertension, heart attack, chronic lung disease, stroke, diabetes, bladder disease, nephrolith, visual problems, hearing problems, and hemorrhoids.
Self-Reported Chronic Medical Conditions | 9 months
  Participants will report whether or not they currently have a list of chronic medical conditions, including but not limited to arthritis, hypertension, heart attack, chronic lung disease, stroke, diabetes, bladder disease, nephrolith, visual problems, hearing problems, and hemorrhoids.
The Chinese version of the Satisfaction with Life Scale | Baseline
  The Chinese version of the Satisfaction with Life Scale will assess the participants' well-being in terms of satisfaction and fulfillment of their current state. Participants will indicate agreement with the content of five items on a 4-point scale (1=Strongly disagree, 4=Strongly agree). Scores will be calculated by summing across the items (range=5-20).
The Chinese version of the Satisfaction with Life Scale | 3 months
  The Chinese version of the Satisfaction with Life Scale will assess the participants' well-being in terms of satisfaction and fulfillment of their current state. Participants will indicate agreement with the content of five items on a 4-point scale (1=Strongly disagree, 4=Strongly agree). Scores will be calculated by summing across the items (range=5-20).
The Chinese version of the Satisfaction with Life Scale | 9 months
  The Chinese version of the Satisfaction with Life Scale will assess the participants' well-being in terms of satisfaction and fulfillment of their current state. Participants will indicate agreement with the content of five items on a 4-point scale (1=Strongly disagree, 4=Strongly agree). Scores will be calculated by summing across the items (range=5-20).
The Chinese version of the nine-item Patient Health Questionnaire | Baseline
  The Chinese version of the nine-item Patient Health Questionnaire will be used to assess the depressive symptoms of the participants over the past two weeks on a 4-point scale (0=Not at all, 1=On several days, 2=More than half the days, 3=Nearly every day). Higher scores indicate a higher level of depressive symptoms (range=0-27).
The Chinese version of the nine-item Patient Health Questionnaire | 3 months
  The Chinese version of the nine-item Patient Health Questionnaire will be used to assess the depressive symptoms of the participants over the past two weeks on a 4-point scale (0=Not at all, 1=On several days, 2=More than half the days, 3=Nearly every day). Higher scores indicate a higher level of depressive symptoms (range=0-27).
The Chinese version of the nine-item Patient Health Questionnaire | 9 months
  The Chinese version of the nine-item Patient Health Questionnaire will be used to assess the depressive symptoms of the participants over the past two weeks on a 4-point scale (0=Not at all, 1=On several days, 2=More than half the days, 3=Nearly every day). Higher scores indicate a higher level of depressive symptoms (range=0-27).
Eating Behaviour Questionnaire from the EatSmart Restaurant Star+ Campaign | Baseline
  The Eating Behaviours questionnaire is an assessment tool adapted from the EatSmart Restaurant Star+ Campaign, an initiative launched by the Department of Health in Hong Kong to promote healthy eating habits. The questionnaire focuses on various aspects of eating behaviors, such as the frequency of cooking at home, dining out, and the consumption patterns of different food groups, including red meat, white meat, fruits, and vegetables.
Eating Behaviour Questionnaire from the EatSmart Restaurant Star+ Campaign | 3 months
  The Eating Behaviours questionnaire is an assessment tool adapted from the EatSmart Restaurant Star+ Campaign, an initiative launched by the Department of Health in Hong Kong to promote healthy eating habits. The questionnaire focuses on various aspects of eating behaviors, such as the frequency of cooking at home, dining out, and the consumption patterns of different food groups, including red meat, white meat, fruits, and vegetables.
Eating Behaviour Questionnaire from the EatSmart Restaurant Star+ Campaign | 9 months
  The Eating Behaviours questionnaire is an assessment tool adapted from the EatSmart Restaurant Star+ Campaign, an initiative launched by the Department of Health in Hong Kong to promote healthy eating habits. The questionnaire focuses on various aspects of eating behaviors, such as the frequency of cooking at home, dining out, and the consumption patterns of different food groups, including red meat, white meat, fruits, and vegetables.

CONTACTS AND LOCATIONS:
Overall Officials: Che Hin Chetwyn Chan, PhD, Principal Investigator — The Education University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Eastern District Health Centre Express, North Point
  - Central and Western District Health Centre Express, Sai Ying Pun
  - Sha Tin District Health Centre Express, Shatin

IPD SHARING:
Plan to Share IPD: No
The collected data, such as weight and height, blood pressure and eating behaviours, may be perceived as sensitive by participants. Further, participants are not informed about sharing their information to parties other than the project team and Hong Kong Society of Rehabilitation.